CLINICAL TRIAL: NCT02042079
Title: Endoscopic Full Thickness Resection With Laparoscopic Assistance, Single Center Single Arm Study
Brief Title: Endoscopic Full Thickness Resection With Laparoscopic Assistance
Acronym: EFTR-LA
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Chan Gyoo Kim, Senior Scientist, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-604
Record Dates: First submitted 2014-01-19; First posted 2014-01-22 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Gastric Subepithelial Tumor
Keywords: Endoscopic full-thickness resection; gastric subepithelial tumor; hybrid-NOTES

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EFTR with LA (Experimental): (Endoscopic full-thickness resection with laparoscopic assistance)
  Interventions: Procedure: EFTR with LA

INTERVENTIONS:
Procedure: EFTR with LA — (Endoscopic full-thickness resection with laparoscopic assistance)

SUMMARY:
The purpose of this study is to evaluate the feasibility of endoscopic full-thickness resection with laparoscopic assistance.

DETAILED DESCRIPTION:
The laparoscopic resection with a linear stapler for subepithelial tumors (SET) can lead to excessive resection of healthy tissue of the gastric wall resulting in deformity or stenosis. Attaining a positive surgical margin is also possible. Endoscopic full-thickness resection (EFTR) can be used for tumor resection by direct visualization of the tumor from inside the stomach lumen leading to a free surgical margin with little resection of healthy tissue. In order to overcome current endoscopic technical limitations, we will combine the conventional laparoscopic approach with EFTR.

ELIGIBILITY:
Inclusion Criteria:

* Gastric subepithelial tumor
* Invasion of muscularis propria on Endoscopic ultrasound
* Tumor size 1.5cm-5cm or increasing size during follow-up

Exclusion Criteria:

* Bleeding tendency,
* Inappropriate condition for surgery with general anesthesia
* Refuse to be enrolled to study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
En-bloc resection and successful closure | 3 months after surgery
  successful En-bloc resection of subepithelial tumor and successful closure of resection site by Endoscopic full-thickness resection with laparoscopic assistance.

SECONDARY OUTCOMES:
number of troche | during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Chan G Kim, M.D., Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea